CLINICAL TRIAL: NCT02432872
Title: A Multicenter，Open-label，Radonmized Study on the Treatment of Older Adult Acute Myeloid Leukemia Patients Aged 55 to 65 Years Old
Brief Title: Treatment of Older Adult Acute Myeloid Leukemia Patients Aged 55 to 65 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianxiang Wang (Unknown)
Responsible Party: Sponsor-Investigator, Jianxiang Wang, vise-president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2015002
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- escalated daunorubicin (Experimental): Daumorubicin 60mg/m2 per day for 3 days combined with Cytaruabine 100mg/m2 per day for 7 days.
  Interventions: Drug: Daunorubicin; Drug: Cytarabine
- standard daunorubicin (Active Comparator): Daunorubicin 45mg/m2 per day for 3 days combined with Cytaruabine 100mg/m2 per day for 7 days.
  Interventions: Drug: Daunorubicin; Drug: Cytarabine
- medium dosage cytarabine (Experimental): 1g/m2 q12h for 3 days as consolidation therapy.
  Interventions: Drug: Cytarabine
- standard dosage cytarabine (Active Comparator): 100mg/m2 cytarabine for 6 days combined with aclacinomycin 20mg per day for 6 days as consolidation therapy.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Daunorubicin — defferent doses of daunorubicin,that is 60mg/m2 for 3 doses compared with 45mg/m2 for 3 doses
  Other Names: daunomycin
  Arms: escalated daunorubicin; standard daunorubicin
Drug: Cytarabine — medium dosage cytarabine（1 g/m2 q12h for 3 days) compared with standard dosage cytarabine(100mg/m2 per day for 6 days)combinated with aclacinomycin（20mg per day for 6 days）for consolidation therapy.
  Other Names: cytosine arabinoside

SUMMARY:
The purpose of this study is to determine whether the escalation dosage of Daunorubicin and cytarabine is effective and safety in the treatment of older adult Chinese acute myeloid leukemia（AML） patients aged 55 to 65 years.

DETAILED DESCRIPTION:
the DA 3+7 regimen is the standard therapy in the AML treatment.Escalated dosage of daunorubicin in induction therapy is reported effective and result in a more rapid response and a higher response rate than does the conventional dose, without additional toxic effects in elderly AML patients between 60 to 65 years.Higher Overall survival rate and Event-free survival rate was obtained in escalated group compared with conventional dose. We are wondering if Chinese older AML patients can benefit from this escalated induction regimen.

High dose cytarabine in AML consolidation is reported improving the survival of elderly AML patients than the conventional dose，but it is not determined in Chinese older adult AML patients.

ELIGIBILITY:
Inclusion Criteria:

* primary AML（except APL patients）;
* ECOG PS:0-2

Exclusion Criteria:

* AML patient who has already received induction treatment, no matter what the outcome is;
* Treatment-related AML;
* Active cancer patients who's condition need to be treated;
* The one with serious infectious diseases（eg.uncontrolled tuberculosis or invasive pulmonary aspergillosis）
* Active heart disease.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
complete remission rate | 2 months
relapse free survival | 3 years
complete remission rate in different risk group | 2 month
treatment-related mortality | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — ChineseAMS
Locations (1):
- Treatment and Diagnosis Center of Leukemia, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided